CLINICAL TRIAL: NCT07083128
Title: Temporal Changes in Parasternal Intercostal Muscle Thickening as a Possible Biomarker for Successful Weaning From Mechanical Ventilation: a Prospective Observational Study
Brief Title: Temporal Change in Parasternal Thickening Fraction as a Predictor for Weaning
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Other Study IDs: Temporal change in PIC
Record Dates: First submitted 2025-07-05; First posted 2025-07-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Weaning From Mechanical Ventilation; Weaning Failure
Keywords: Parasternal thickening; failed weaning; extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Parasternal intercostal thickening — Temporal change in parasternal intercostal thickening fraction at initiation and 30 minutes of spontaneous breathing trial

SUMMARY:
optimal time to liberate from mechanical ventilation is highly prioritized since improper extubation time lead to serious consequences

DETAILED DESCRIPTION:
Several parameters were proposed to assess proper weaning time including diaphragmatic ultrasound and extra-diaghragmatic muscles. previous research concluded an ability of parasternal intercostal (PIC) thickening to predict weaning outcomes. researchers of current study assumed that temporal changes in PIC thickening would provide greater ability to predict weaning outcomes

ELIGIBILITY:
Inclusion Criteria:

- Mechanically ventilated for 24 hours or more ready for weaning

Exclusion Criteria:

* Refusal Tracheostomized Inability to obtain ultrasound views patients with neuromuscular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient who are mechanically ventilated for 24 hours or more and ready for weaning
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of change in PIC-TF in predicting successful weaning from mechanical ventilation | At baseline and 30 minutes after initiation of spontaneous breathing trial
  percentage of change in PIC TF in predicting weaning outcome

SECONDARY OUTCOMES:
Accuracy of change in PIC-TF to predict reintubation | At baseline and 30 minutes after initiation of spontaneous breathing trial
  percentage of change in PIC TF at start and end of spontaneous breathing trial

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shared due to confidentiality, legal constraints, or the need to protect intellectual property rights.

REFERENCES:
- [Result] Helmy MA, Hasanin A, Milad LM, Mostafa M, Hamimy WI, Muhareb RS, Raafat H. Ability of parasternal intercostal muscle thickening fraction to predict reintubation in surgical patients with sepsis. BMC Anesthesiol. 2024 Aug 22;24(1):294. doi: 10.1186/s12871-024-02666-8. PMID 39174907
- [Result] Helmy MA, Milad LM, Hasanin AM, Mostafa M, Mannaa AH, Youssef MM, Abdelaziz M, Alkonaiesy R, Elshal MM, Hosny O. Parasternal intercostal thickening at hospital admission: a promising indicator for mechanical ventilation risk in subjects with severe COVID-19. J Clin Monit Comput. 2023 Oct;37(5):1287-1293. doi: 10.1007/s10877-023-00989-4. Epub 2023 Mar 24. PMID 36961635
- [Result] Helmy MA, Hasanin A, Milad LM, Mostafa M, Fathy S. Parasternal intercostal muscle thickening as a predictor of non-invasive ventilation failure in patients with COVID-19. Anaesth Crit Care Pain Med. 2022 Jun;41(3):101063. doi: 10.1016/j.accpm.2022.101063. Epub 2022 Apr 26. No abstract available. PMID 35487407
- [Result] Helmy MA, Magdy Milad L, Osman SH, Ali MA, Hasanin A. Diaphragmatic excursion: A possible key player for predicting successful weaning in patients with severe COVID-19. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100875. doi: 10.1016/j.accpm.2021.100875. Epub 2021 Apr 30. No abstract available. PMID 33940248
- [Result] Adolf Helmy M, Magdy Milad L, Hasanin A, Mostafa M. The novel use of diaphragmatic excursion on hospital admission to predict the need for ventilatory support in patients with coronavirus disease 2019. Anaesth Crit Care Pain Med. 2021 Dec;40(6):100976. doi: 10.1016/j.accpm.2021.100976. Epub 2021 Nov 5. PMID 34748940